CLINICAL TRIAL: NCT03481218
Title: Quality of Life and Personality Traits in Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: MN-2017
Record Dates: First submitted 2018-03-13; First posted 2018-03-29 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Type 1 Diabetes; Quality of Life
Keywords: Type 1 diabetes; Quality of life; Personality traits; Young adults
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 1 diabetes: Young adults (male and female) between the ages of 18 and 35, who have type 1 diabetes for at least one year.
  Interventions: Other: The World Health Organization Quality of Life (WHOQOL) -BREF; Other: The Satisfaction With Life Scale - SWLS; Other: Big Five Inventory - BFI; John in Srivastava, 1999
- Individuals without chronic diseases: Young adults (male and female) between the ages of 18 and 35, without chronic diseases.
  Interventions: Other: The World Health Organization Quality of Life (WHOQOL) -BREF; Other: The Satisfaction With Life Scale - SWLS

INTERVENTIONS:
Other: The World Health Organization Quality of Life (WHOQOL) -BREF — The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment.
Other: The Satisfaction With Life Scale - SWLS — The SWLS is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life.
Other: Big Five Inventory - BFI; John in Srivastava, 1999 — The Big Five Inventory (BFI) is a self-report inventory designed to measure the Big Five dimensions.
  Groups: Patients with type 1 diabetes

SUMMARY:
The aims of this study are to examine the differences in the quality of life among individuals with type 1 diabetes and individuals without chronic diseases, differences in the quality of life among men and women with type 1 diabetes and the differences in the quality of life among individuals with good and poor glycaemic control. The relationship between personality traits and the management of disease in patients with type 1 diabetes will also be examined.

DETAILED DESCRIPTION:
Diabetes affects the daily life of patients, chronic diseases have a major impact on the quality of life of individuals. Chronic illness affects family life of an individual, his professional life, as well as leisure activities, chronic illness can also increase worries, fears, feelings of sadness and helplessness.

Past studies examining the quality of life construct in patients with type 1 diabetes (T1D) showed that patients achieved lower levels of life quality, compared to individuals without T1D. Studies show that women with T1D achieve lower scores on the quality of life scales than men with T1D and differences in gender are already present in adolescence.

Patients with poor glycaemic control achieve lower results on the quality of life scales, the effect of hemoglobin on the quality of life is direct, as well as indirect.

The studies in which they examined the attitudes of personality traits with diabetes management show that two personality traits are associated with the management of the disease, the successful management of the disease is primarily associated with the conscientiousness. Concerning the effect of neuroticism on the management of the disease, research results are contradictory.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35
* Diagnosed with Type 1 diabetes for at least one year (for the T1D group)
* Willing to participate in study

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Young adults of 18 to 35 years of age with type 1 diabetes and young adults of 18 to 35 years of age without chronic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Differences in quality of life | 15 minutes
  Differences in quality of life in patients with T1D and individuals without chronic diseases. Quality of life will be measured with the WHOQOL-BREF quality of life assessment tool (questionnaire).
Personality traits associated with diabetes management | 15 minutes
  Which personality traits are associated with good and poor diabetes management. Personality traits will be measured with The Big Five Inventory questionnaire.

SECONDARY OUTCOMES:
Differences in quality of life based on gender | 15 minutes
  Differences in quality of life between men and women with T1D. Quality of life will be measured with the WHOQOL-BREF quality of life assessment tool (questionnaire).
Differences in quality of life based on glycaemic control | 15 minutes
  Differences in quality of life between patients with good and bad glycaemic control. Quality of life will be measured with the WHOQOL-BREF quality of life assessment tool (questionnaire). Glycaemic control will be reported from participants (HbA1c).

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - University Children's Hospital Ljubljana, Ljubljana, Slovenija/Osrednja Regija
  - University of Ljubljana, Faculty of Arts, Department of psychology, Ljubljana, Slovenija/Osrednja Regija

REFERENCES:
- [Background] Alvarado-Martel D, Velasco R, Sanchez-Hernandez RM, Carrillo A, Novoa FJ, Wagner AM. Quality of life and type 1 diabetes: a study assessing patients' perceptions and self-management needs. Patient Prefer Adherence. 2015 Sep 14;9:1315-23. doi: 10.2147/PPA.S87310. eCollection 2015. PMID 26396503
- [Background] Booth-Kewley S, Vickers RR Jr. Associations between major domains of personality and health behavior. J Pers. 1994 Sep;62(3):281-98. doi: 10.1111/j.1467-6494.1994.tb00298.x. PMID 7965560
- [Background] Hilliard ME, Mann KA, Peugh JL, Hood KK. How poorer quality of life in adolescence predicts subsequent type 1 diabetes management and control. Patient Educ Couns. 2013 Apr;91(1):120-5. doi: 10.1016/j.pec.2012.10.014. Epub 2012 Nov 22. PMID 23182614
- [Background] Lawrence JM, Yi-Frazier JP, Black MH, Anderson A, Hood K, Imperatore G, Klingensmith GJ, Naughton M, Mayer-Davis EJ, Seid M; SEARCH for Diabetes in Youth Study Group. Demographic and clinical correlates of diabetes-related quality of life among youth with type 1 diabetes. J Pediatr. 2012 Aug;161(2):201-7.e2. doi: 10.1016/j.jpeds.2012.01.016. Epub 2012 Feb 22. PMID 22361221
- [Background] Lane JD, McCaskill CC, Williams PG, Parekh PI, Feinglos MN, Surwit RS. Personality correlates of glycemic control in type 2 diabetes. Diabetes Care. 2000 Sep;23(9):1321-5. doi: 10.2337/diacare.23.9.1321. PMID 10977026
- [Background] Majumder E, Cogen FR, Monaghan M. Self-Management Strategies in Emerging Adults With Type 1 Diabetes. J Pediatr Health Care. 2017 Jan-Feb;31(1):29-36. doi: 10.1016/j.pedhc.2016.01.003. Epub 2016 Feb 6. PMID 26861574
- [Background] Martyn-Nemeth P, Quinn L, Penckofer S, Park C, Hofer V, Burke L. Fear of hypoglycemia: Influence on glycemic variability and self-management behavior in young adults with type 1 diabetes. J Diabetes Complications. 2017 Apr;31(4):735-741. doi: 10.1016/j.jdiacomp.2016.12.015. Epub 2017 Jan 20. PMID 28143733
- [Background] Naughton MJ, Yi-Frazier JP, Morgan TM, Seid M, Lawrence JM, Klingensmith GJ, Waitzfelder B, Standiford DA, Loots B; SEARCH for Diabetes in Youth Study Group. Longitudinal associations between sex, diabetes self-care, and health-related quality of life among youth with type 1 or type 2 diabetes mellitus. J Pediatr. 2014 Jun;164(6):1376-83.e1. doi: 10.1016/j.jpeds.2014.01.027. Epub 2014 Feb 26. PMID 24582483
- [Background] Nielsen HB, Ovesen LL, Mortensen LH, Lau CJ, Joensen LE. Type 1 diabetes, quality of life, occupational status and education level - A comparative population-based study. Diabetes Res Clin Pract. 2016 Nov;121:62-68. doi: 10.1016/j.diabres.2016.08.021. Epub 2016 Sep 8. PMID 27662040
- [Background] Rassart J, Luyckx K, Moons P, Weets I. Personality and self-esteem in emerging adults with Type 1 diabetes. J Psychosom Res. 2014 Feb;76(2):139-45. doi: 10.1016/j.jpsychores.2013.11.015. Epub 2013 Dec 6. PMID 24439690
- [Background] Rassart J, Luyckx K, Klimstra TA, Moons P, Groven C, Weets I. Personality and illness adaptation in adults with type 1 diabetes: the intervening role of illness coping and perceptions. J Clin Psychol Med Settings. 2014 Mar;21(1):41-55. doi: 10.1007/s10880-014-9387-2. PMID 24496583
- [Background] Raynor DA, Levine H. Associations between the five-factor model of personality and health behaviors among college students. J Am Coll Health. 2009 Jul-Aug;58(1):73-81. doi: 10.3200/JACH.58.1.73-82. PMID 19592356
- [Background] Rechenberg K, Whittemore R, Grey M. Anxiety in Youth With Type 1 Diabetes. J Pediatr Nurs. 2017 Jan-Feb;32:64-71. doi: 10.1016/j.pedn.2016.08.007. Epub 2016 Sep 20. PMID 27663096
- [Background] Strandberg RB, Graue M, Wentzel-Larsen T, Peyrot M, Wahl AK, Rokne B. The relationships among fear of hypoglycaemia, diabetes-related quality of life and psychological well-being in Norwegian adults with Type 1 diabetes. Diabetes Res Clin Pract. 2017 Feb;124:11-19. doi: 10.1016/j.diabres.2016.12.018. Epub 2016 Dec 27. PMID 28081448
- [Background] Trento M, Panero F, Porta M, Gruden G, Barutta F, Cerutti F, Gambino R, Perotto M, Cavallo Perin P, Bruno G; Piedmont Study Group for Diabetes Epidemiology. Diabetes-specific variables associated with quality of life changes in young diabetic people: the type 1 diabetes Registry of Turin (Italy). Nutr Metab Cardiovasc Dis. 2013 Oct;23(10):1031-6. doi: 10.1016/j.numecd.2013.01.004. Epub 2013 Mar 7. PMID 23466181
- [Background] Wheeler K, Wagaman A, McCord D. Personality traits as predictors of adherence in adolescents with type I diabetes. J Child Adolesc Psychiatr Nurs. 2012 May;25(2):66-74. doi: 10.1111/j.1744-6171.2012.00329.x. PMID 22512523